CLINICAL TRIAL: NCT03112096
Title: A Phase I [18F]THK-5351 Positron Emission Computed Tomography Study of Biodistribution, Pharmacokinetics and Safety in Cognitively Healthy Subjects and Patients With Alzheimer's Disease
Brief Title: A Phase I [18F]THK-5351 Positron Emission Tomography Study in Healthy Subjects and Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: THK-15001
Record Dates: First submitted 2017-03-26; First posted 2017-04-13 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Alzheimer Disease
Keywords: Tau; neurodegeneration; positron emission tomography
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain; Nerve Degeneration | interventions — THK5351

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitively Healthy Subjects (Experimental): Cognitively healthy subjects will receive an IV injection, [18F]THK-5351 injection
  Interventions: Drug: [18F]THK-5351
- Alzheimer's Disease Subjects (Experimental): Cognitively healthy subjects will receive an IV injection, [18F]THK-5351 injection
  Interventions: Drug: [18F]THK-5351

INTERVENTIONS:
Drug: [18F]THK-5351 — Imaging for evaluating the biodistribution, pharmacokinetics and safety of abnormal tau protein in the brain
  Other Names: FluoroTau

SUMMARY:
This is a study to evaluate biodistribution, pharmacokinetics and safety of [18F]THK-5351 positron emission computed tomography in Cognitively Healthy Subjects and Patients with Alzheimer's Disease.

DETAILED DESCRIPTION:
This is a study to evaluate biodistribution, pharmacokinetics and safety of [18F]THK-5351 positron emission computed tomography. Ten cognitively healthy subjects and 10 patients with Alzheimer's Disease will be enrolled. The primary outcome measures are to evaluate pharmacokinetics of [18F]THK-5351 Positron Emission Tomography imaging . Tracer biodistribution will be evaluated by global and regional standardized uptake value ratio of [18F]THK-5351 in the brain. Safety. For safety assessment, a physical examination, Electrocardiogram and vital signs will be performed at baseline and at the completion of all imaging to assess for interval change.

ELIGIBILITY:
Inclusion Criteria;

- General Subject Inclusion Criteria

In order to be eligible for participation in this trial, the subject must:

1. Be able to read at a 6th grade level or equivalent, (as determined by the investigator, and must have a history of academic achievement and/or employment sufficient to exclude mental retardation.)
2. Be able to speak, read, hear, and understand the language of the trial staff, and the informed consent form, and possess the ability to respond verbally to questions, follow instructions, and complete questionnaires and detailed neuropsychological test.
3. Have results of clinical laboratory tests/physical examination, vital signs, and Electrocardiogram within normal limits (at 45 days prior to [18F]THK-5351 Positron Emission Tomography scan ) or clinically acceptable to the investigator at screening.
4. Be able to possess the ability to respond verbally to questions, follow instructions, and underwent research assessment, including brain images based on the investigator's judgment. Each subject is also able and willing to adhere visit schedules.
5. If female, not be of childbearing potential as indicated by one of the following

   1. has reached natural menopause, defined as ≥ 24 months of spontaneous amenorrhea or
   2. has had a hysterectomy; or
   3. has had a bilateral oophorectomy (with or without a hysterectomy) and more than 6 weeks have passed since the surgery.
6. Each subject (or legal representative) must sign the informed consent form in accordance with local requirements after the scope and nature of the investigation have been explained to them, and before screening assessments.

   - Normal Subject Inclusion Criteria

<!-- -->

1. . Be ≥ 20 years of age at the screening visit
2. Each subject must not report a history of memory decline with gradual onset and slow progression, that is either corroborated by an informant who knows the subject well or is documented in medical records. Each subject must have general cognitive function and activities of daily living sufficiently intact, based on clinical assessment, so as not to meet criteria for mild AD dementia (based on DSM-IV-TR(Diagnostic and Statistical Manual of Mental Disorders, 4th Edition) and NINCDS-ADRDA(National Institute of Neurological and Communicative Disorders and Stroke; Alzheimer's Disease and Related Disorders Association) criteria).
3. Each subject must have results of Korean-Mini Mental State Exam (K-MMSE) at screening that is ≥1.5 SD above the appropriate population mean, corrected age and education.
4. Each subject must not have objective impairment in memory at screening that is ≥1.5 SD above the appropriate population mean, corrected age and education, as measured by the Seoul Verbal Learning Test (SVLT) delayed recall score of the Seoul Neuropsychological Screening Battery (SNSB)-Ⅱ.
5. Each subject must have normal level of general cognitive function and activities of daily living sufficiently intact, that is 0 score as measured by the Clinical Dementia Rating (CDR).
6. Each subject must have an MRI scan obtained at screening that supports diagnosing the current status of normal cognition. The MRI for research must be consistent and sufficient in quality enough to analyze volume of interest (VOI) with partial volume correction (Detailed protocol is described in the MRI scanning manual).
7. Each subject must be willing to provided blood samples for genotyping apolipoprotein E.

   * Alzheimer's Disease Inclusion Criteria

<!-- -->

1. Be ≥ 50 and < 80 years of age at the Screening Visit.
2. Each subject must have general cognitive function and activities of daily living impairment, based on clinical assessment, so as to meet criteria for AD dementia (based on DSM-IV-TR and NINCDS-ADRDA criteria).
3. Each subject's K-MMSE score ranges 15-26 and CDR 0.5, 1 or 2.
4. Each subject must have a Rosen-modified Hachinski Ischemia Score ≤ 4 at Screening.
5. Each subject must have a reliable and competent trial partner/informant who must have a close relationship with the subject, and can be accompanied at all visits in this study.
6. Each subject must have an MRI scan obtained at screening that supports diagnosing Alzheimer's disease. The MRI for research must be consistent and sufficient in quality enough to analyze volume of interest (VOI) with partial volume correction (Detailed protocol is described in the MRI scanning manual).
7. If receiving some medications, be on a stable dose for at least the 4 weeks before performing THK5351 PET scan, and the subject must be willing to remain on the same dose for the duration of the trial.
8. Each subject must be willing to provided blood samples for genotyping ApoE.
9. Each subject must shows positive in amyloid PET scan.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject fulfil any single criteria described below:

* General Exclusion Criteria 1. Based on the investigators' judgement, if the patient is not capable of communicating with the site personnel, if the patient is not proficient in the language in which the psychometric tests will be completed, or if the patient is not sufficient for compliance with the study procedures.

  2. The patient has an abnormal physical examination, abnormal laboratory test or electrocardiography results at the screening that are clinically significant to affect results of the research, as judged by the investigator.

  3. If the patient has or is suspicious of having a hypersensitivity or allergy to [18F] THK-5351 or its derivatives.

  4. The patient is pregnant, is attempting to become pregnant, or is nursing (breast-feeding) children.

  5. The patient has a history of alcoholism or drug dependency/abuse within the last 2 years before screening.

  6. The patient has contraindications to undergo PET or MRI, which include but are not restricted to the examples below: claustrophobia, cardiac pacemaker, metal devices around the eye or spinal cord, cochlear implant, etc.) at the screening visit.

  7. The patient has been treated with any investigational medicinal product (IMP) within 30 days prior to the screening visit.

  8. The patient has been tested positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), HIV Antibody, or syphilis serum test at the screening visit.

  9. The patient has been receiving an anti-cholinergic drug in a regular basis within 3 months prior to the screening visit.

  10. The patient has evidence of a clinically relevant neurological disorders other than the disease being studied (i.e., prodromal AD) at screening, including but not limited to: territorial cerebral infarction, intracranial hemorrhage, multiple sclerosis, neurosyphilis, mental retardation, hypoxic encephalopathy, major head trauma with loss of consciousness that led to persistent cognitive deficits.

  11. The patients has disorders related to blood coagulation which could be inappropriate for arterial or venous sampling.
* Normal Subject Exclusion Criteria 1. The patient has evidence of a clinically significant medical disorder, neurological disorder, has an abnormal physical examination or abnormal laboratory evaluations from the screening visit, or has other abnormal findings that are clinically significant, as judged by the investigator.

  2. The patient has more than one direct family members who were diagnosed with Alzheimer's disease.
* Alzheimer's Disease Exclusion Criteria

  1. The patient has evidence of any clinically significant neurodegenerative disease, or other serious neurological disorders other than AD including but not limited to stroke, traumatic brain injury, non-Alzheimer tauopathy, Parkinson's disease, or has evidence of a clinically relevant or unstable psychiatric disorders, including but not limited to major depression, schizophrenia, or bipolar disorder.
  2. The patient has more than two direct family members who were diagnosed with Alzheimer's disease.
  3. The patient has a stroke or an evidence of significant cerebrovascular disease from screening imaging scan that is clinically important in the investigator's opinion.
  4. The patient has received any of the treatments targeting tau protein prior to [18F]THK-5351 PET scan.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum Serum Concentration (Cmax) of [18F]THK-5351 | 0-90 minutes post injection
  Compare time activity curve and calculate maximum serum concentration (Cmax) of each region of interest of [18F]THK-5351 positron emission computed tomography in cognitively healthy subjects and patients with Alzheimer's disease
Assess global and regional tau deposition as measured by standard uptake value ratio (SUVR) of [18F]THK-5351 | 0-90 minutes post injection or 50-70 minutes post injection
  Compare Standard uptake value ratio (SUVR) and distribution of [18F]THK-5351 in cognitively healthy subjects and patients with Alzheimer's disease

SECONDARY OUTCOMES:
Correlation between standard uptake value ratio (SUVR) and distribution volume of ratio(DVR) of [18F]THK-5351 positron emission computed tomography | 0-90 minutes post injection or 50-70 minutes post injection
  We will evaluate correlation between standard uptake value ratio (SUVR) and distribution volume of ratio(DVR) of[18F]THK-5351 positron emission computed tomography
Optimal scanning time for brain imaging using F-18 THK-5351. | 0-90 minutes post injection
  PET data will be acquired during a 90-min dynamic brain PET scan and will be started simultaneously with the injection of 10mCi of F-18 THK-5351. Reconstruction of PET imaging with several time frame will be compared.
Concentrations of metabolite in plasma of [18F]THK-5351 | 0-90 minutes post injection or 50-70 minutes post injection
  Plasma metabolite concentrations [18F]THK-5351 will be assessed.
Number of participants with treatment related adverse events as a measure of safety | 0-90 minutes post injection or 50-70 minutes post injection
  For safety assessment, a physical examination, EKG and vital signs will be performed at baseline and at the completion of all imaging to assess for interval change.

CONTACTS AND LOCATIONS:
Overall Officials: JaeEun Kim, Study Director — Asan Foundation
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided